CLINICAL TRIAL: NCT03146143
Title: Effect of Ultra Filtration on Extravascular Lung Water Assessed by Lung Ultrasound in Pediatric Cardiac Surgery
Brief Title: Ultrafiltration Effect on Extravascular Lung Water in Pediatric Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Elayashy Mohamed Ahmed Hassan, clinical professor, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N-19-2017
Record Dates: First submitted 2017-04-29; First posted 2017-05-09 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Congenital Cardiac Disorders
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Ultrafiltration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrafiltration group (Experimental): ultrafiltration after cardiopulmonary bypass in congenital cardiac surgery
  Interventions: Procedure: ultrafiltration
- non ultrafiltration control group (No Intervention): no ultrafiltration will be applied in this group

INTERVENTIONS:
Procedure: ultrafiltration — ultrafiltration after cardiopulmonary bypass
  Arms: ultrafiltration group

SUMMARY:
study will assess the effect the ultrafiltration after pediatric congenital heart surgery on cardiopulmonary bypass. patients will be divided into two groups. first group will receive ultrafiltration and the second group will be control group without filtration.

we will assess extravascular lung water by lung ultrasound, arterial oxygen tension and duration of ventilation.

DETAILED DESCRIPTION:
The anesthesiologist will interview the guardians; examine the patients, checking all routine investigations include: CBC(complete blood count), coagulation profile, liver function tests, renal function tests, blood grouping, chest X-ray, recent echocardiography and angiography if available.

Children will be received Midazolam 0.3 mg/kg IM (intramuscular) and Atropine 0.02 mg/kg IM 10 min as pre-medication before induction.

Induction of anesthesia will be established using fentanyl, 1-5µg/kg, ketamine 1-2 g/kg. Atracurium 0.5mg/kg will be administered to facilitate endotracheal intubation and repeated intraoperative as required to maintain muscle relaxation. Anesthesia will be maintained using sevoflurane 0.3%-2 % in oxygen-air mixture (1:1 ratio). A central venous line will be inserted and arterial line for invasive blood pressure monitoring. The use of inotropes will be guided by the patient's hemodynamics after surgical repair. Dobutamine 5-10 µg/Kg/min, Tridil 1-4 µg/Kg/ min, Adrenaline 0.05µg/kg/min or Milrinone 0.5µg/kg/min will be used according to pathophysiology and Intraoperative state of patient.

In all patients, a median sternotomy will be performed. CPB will be initiated after full heparinization in a dose of 300-400 I.U to achieve a n ACT( activated clotting time) of 450 sec or 3 times baseline reading followed by the standard aorta-bicaval cannulation. A membrane oxygenator (Mini-max Plus; Medtronic Inc., Anaheim, CA) and a non-pulsatile roller pump (model 10.10.00; Stôckert Instruments; Munich, Germany) will be used. Venting of the left heart will be performed with a left atrial vent inserted through a small incision at the interatrial septum. Priming fluids consist of lactated Ringer's solution supplemented with heparin. Fresh whole blood was added to the priming solution in appropriate amounts to achieve a hematocrit of 20% to 22% during CPB ( cardiopulmonary bypass). Moderate hypothermia (26°C to 28°C) will be used during CPB.

After cardiac repair the patient will be weaned from CPB. protamine will be given 3-4 mg/kg to reverse heparin. The control group will not subjected to ultrafiltration and the ultrafiltration group will be subjected to conventional ultrafiltration guided by hematocrit level 28%.

Blood transfusion on bypass will be guided by hemoglobin level in ABG (arterial blood gases) to keep HB% (hemoglobin) above 7mg/dl. Transfusion of blood products will be guided by clinical state of patient.

Assessment of extra vascular lung water busing lung ultrasound. Lung ultrasound will be performed to diagnose EVLW (extravascular lung water). A M. turbo sonosite ultrasound system with pediatric linear probe (frequency 13-6 MHz( megahertz); Fujifilm, sonosite, inc. USA) will be used. Chest ultrasound will be performed using the 12 reg ions method. Intercostals spaces on each side will be examined anteriorly (midclavicular line), laterally (anterior axillary line) and posteriorly (posterior axillary line) (2).

Four ultrasound aeration patterns: a. Normal aeration (N): 0 score ; line sliding sign associated with respiratory movement or less than 3 B lines ; b. Moderate loss of lung aeration: score 1 ; a clear number of multiple visible B-lines with horizontal spacing between adjacent B lines ≤ 7 mm (B7 lines) c. Severe loss of lung aeration: score 2; multiple B lines fused together that were difficult to count with horizontal spacing between adjacent B lines ≤ 3 mm (B3 lines); and d. Pulmonary consolidation: score 3; hypoechoic lung tissue, accompanied by dynamic air bronchogram.

The final LUS (lung ultrasound score) of the patient was the sum of each regional ultrasound score (ranging from 0 to 36).

The lung ultrasound score will be recorded at baseline and at end of surgery. ABGs will be taken to measure p/f ratio. Hemodynamic (HR and MAP) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Pediatrics undergoing congenital heart surgery
* Age 1 months to 4 years
* ASA II and III
* Weight more than 3 kg

Exclusion Criteria:

* pre-operative mechanical ventilation
* Pre-operative inotropic support.
* Patients with lung disease (asthma, bronchiectasis)
* Preoperative renal impairment (cr > 1.5mg/dl)

Ages: 1 Month to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2017-10-15 (Actual)

PRIMARY OUTCOMES:
Lung ultrasound score | at the end of surgery
  assess extravascular lung water in the form of B lines in lung ultrasound

SECONDARY OUTCOMES:
lung ultrasound score | baseline 5 minutes after induction of anesthesia
  assess extravascular lung water in the form of B lines in lung ultrasound
ultrafiltration volume | at the end of surgery
urea | baseline, day 1 postoperative in icu. day 2 postoperative in icu
duration of ventilation | up to 2 weeks
creatinine | baseline, day 1 postoperative in icu. day 2 postoperative in icu
P/F ratio | baseline 5 minutes after induction of anesthesia and at the end of surgery
  po2 measured by arterial blood gases and then divided by fio2 to get P/F ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy Hospital , Faculty of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Agricola E, Bove T, Oppizzi M, Marino G, Zangrillo A, Margonato A, Picano E. "Ultrasound comet-tail images": a marker of pulmonary edema: a comparative study with wedge pressure and extravascular lung water. Chest. 2005 May;127(5):1690-5. doi: 10.1378/chest.127.5.1690. PMID 15888847
- [Background] Copetti R, Cattarossi L. Ultrasound diagnosis of pneumonia in children. Radiol Med. 2008 Mar;113(2):190-8. doi: 10.1007/s11547-008-0247-8. Epub 2008 Apr 2. English, Italian. PMID 18386121
- [Background] Zhao Z, Jiang L, Xi X, Jiang Q, Zhu B, Wang M, Xing J, Zhang D. Prognostic value of extravascular lung water assessed with lung ultrasound score by chest sonography in patients with acute respiratory distress syndrome. BMC Pulm Med. 2015 Aug 23;15:98. doi: 10.1186/s12890-015-0091-2. PMID 26298866
- [Derived] Elayashy M, Madkour MA, Mahmoud AAA, Hosny H, Hussein A, Nabih A, Lofty A, Hamza HM, Hassan P, Wagih M, Mohamed AK. Effect of ultrafiltration on extravascular lung water assessed by lung ultrasound in children undergoing cardiac surgery: a randomized prospective study. BMC Anesthesiol. 2019 Jun 4;19(1):93. doi: 10.1186/s12871-019-0771-1. PMID 31159739